CLINICAL TRIAL: NCT06178159
Title: A Phase II, Multicenter, Open-Label Neoadjuvant Study to Evaluate the Safety and Efficacy of Disitamab Vedotin in Combination With Pertuzumab With or Without Toripalimab for HER2 Positive Breast Cancer
Brief Title: DV in Combination With Pertuzumab With or Without Toripalimab Neoadjuvant Therapy With HER2-positive Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC48-C026
Record Dates: First submitted 2023-12-03; First posted 2023-12-20 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; HER2-positive
MeSH Terms: conditions — Breast Neoplasms | interventions — disitamab vedotin; pertuzumab; toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Disitamab Vedotin + Pertuzumab (Experimental): Disitamab Vedotin With Pertuzumab arm
  Interventions: Drug: Disitamab Vedotin Injection; Drug: Pertuzumab Injection
- Disitamab Vedotin + Toripalimab+ Pertuzumab (Experimental): Disitamab Vedotin+ Toripalimab with Pertuzumab arm
  Interventions: Drug: Disitamab Vedotin Injection; Drug: Pertuzumab Injection; Drug: Toripalimab

INTERVENTIONS:
Drug: Disitamab Vedotin Injection — 2.0mg/kg, intravenous infusion，D1, every 2 weeks, Every 6 weeks is a treatment cycle. A total of 3 cycles (18 weeks) of treatment are performed.
  Other Names: DV,RC48-ADC
Drug: Pertuzumab Injection — Initial dose 840mg, after 2nd dose 420mg intravenous infusion， every 3 weeks
Drug: Toripalimab — 3.0 mg/kg, intravenous infusion, D1, every 2 weeks
  Other Names: JS001
  Arms: Disitamab Vedotin + Toripalimab+ Pertuzumab

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Disitamab Vedotin in combination with Pertuzumab with or without Toripalimab neoadjuvant therapy in patients with HER2-positive breast cancer.

DETAILED DESCRIPTION:
This is an open-label, randomized, multicenter, Phase II Study designed to evaluate safety and efficacy of Disitamab Vedotin in combination with Pertuzumab with or without Toripalimab neoadjuvant therapy inr patients with HER2-positive breast cancer.

The primary objectives of the study are to explore combination neoadjuvant therapy in participants with previously untreated HER2-positive breast cancer, by assessment of pCR .

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate and sign the informed consent form;
2. Ages≥18 years;
3. Histopathologically confirmed invasive breast cancer, clinical stage T2-3 (tumor diameter > 2 cm), cN0- 3, M0;
4. Invasive breast tumour tissue confirmed HER2-positive by the central laboratory, defined as HER2 protein expression of IHC 3+ by immunohistochemistry (IHC) or IHC 2+ with amplification by in situ hybridisation (ISH) (according to the HER2 Guidelines for Breast Cancer, 2019 edition); and specimens from the primary site of the tumour for HER2 testing (wax blocks, sections or fresh tissue are acceptable) can be provided for HER2 testing;
5. Subjects who tolerate and are scheduled to undergo radical breast cancer surgery and have not received any prior anti-tumour systemic therapy for breast cancer, as assessed by site.
6. At least one measurable lesion according to RECIST v1.1 criteria;
7. Cardiac function: New York Heart Association (NYHA) class <3; left ventricular ejection fraction ≥55%;
8. Bone marrow or organ function, the following criteria should be met within 7 days prior to study dosing (normal values are based on the clinical trial centre, no transfusion of blood, haematopoietic stimulating factors, albumin or blood products within 14 days prior to the test): haemoglobin ≥ 90 g/L; absolute neutrophil count (ANC) ≥ 1.5 × 109 /L; platelets ≥ 100 × 109 /L; serum total bilirubin ≤ 1.5 times the Upper Limit of Normal (ULN); Albuminous Transaminase (AST) and Albuminous Transaminase (ALT) ≤ 2.5 × ULN; International Normalised Ratio (INR) and Activated Fractional Thromboplastin Time ≤ 1.5 × ULN; and Creatinine Clearance (CrCl) ≥ 50 mL/min according to the Cockcroft-Gault formula method;
9. Subjects of childbearing potential who meet the following criteria:

   1. A serum pregnancy test (minimum sensitivity of 25 mIU/mL or equivalent units of β-human chorionic gonadotropin [β-hCG]) must be negative within 72 hours prior to the first dose of study intervention. Subjects with false-positive results and confirmed non-pregnancy will be eligible for participation in the study.
   2. Must agree to contraception for the duration of the study and for at least 6 months after the last dose of study drug (7 months after the last dose of patulizumab).
   3. Must agree not to breastfeed or donate eggs from the time of signing the informed consent until 6 months after the last dose of study drug (7 months after the last dose of patulizumab).
   4. If sexually active and likely to result in pregnancy, use of at least 2 acceptable contraceptive methods, at least 1 of which must be highly effective, must be continued from the time of informed consent for at least 6 months after the last dose of study drug (7 months after the last dose of patulizumab).
10. Subjects of childbearing potential who meet the following criteria:

    1. Must agree not to donate sperm from the time of signing the informed consent until at least 4 months after the last dose of study drug (7 months after the last dose of patulizumab).
    2. If sexual intercourse with a person of childbearing potential is likely to result in pregnancy, the use of at least 2 acceptable forms of contraception, at least 1 of which must be highly effective, must be continuous, beginning at the time of informed consent and continuing until at least 4 months after the last dose of study drug (7 months after the last dose of patuximab).
    3. If sex with a pregnant or breastfeeding patient, condom use must be continued from the start of informed consent and continue until at least 4 months after the last dose of study drug (7 months after the last dose of patuximab).

12. Be able to understand the requirements of the trial and be willing and able to comply with the trial and follow up procedural arrangements.

Exclusion Criteria:

1. With bilateral invasive breast cancer
2. Previous history of invasive breast cancer
3. Previous carcinoma in situ of the breast with adjuvant endocrine therapy within 5 years of surgery
4. Prior treatment with PD-(L)1, PD-L2, CTLA4 inhibitors and other antibody-coupled drugs
5. Prior anti-HER2 therapy including but not limited to ADC
6. Use of investigational drugs or major surgery within 4 weeks prior to start of study drug administration
7. Vaccination with live or live attenuated vaccine within 4 weeks prior to the start of study drug administration or planned for the duration of the study;
8. History of previous allogeneic haematopoietic stem cell transplantation or organ transplantation;
9. Uncontrolled or significant cardiovascular disease, including (but not limited to): any of the following within 6 months prior to the first dose: e.g., congestive heart failure (NYHA class III or IV), myocardial infarction or cerebral infarction (except for lacunar cerebral infarction), pulmonary embolism, unstable angina, or arrhythmia requiring treatment at screening; primary cardiomyopathy (e.g., dilated cardiomyopathy, Primary cardiomyopathies (e.g., dilated cardiomyopathy, hypertrophic cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy, restrictive cardiomyopathy, indeterminate cardiomyopathy); history of clinically significant prolongation of the QTc period, grade II type II AV block or grade III AV block or QTc interval (F method) >470 msec (women) or >450 msec (men); atrial fibrillation (EHRA grade ≥2b); uncontrolled hypertension that is judged by the investigator to be unsuitable; and Hypertension, judged by the investigator to be unsuitable for participation in the study;
10. History of interstitial lung disease requiring treatment or current severe lung disease including, but not limited to, active tuberculosis, interstitial lung disease;
11. A clear past or present history of a neurological or psychiatric disorder, including epilepsy or dementia;
12. Persistent grade ≥2 sensory or motor neuropathy;
13. Active infection requiring systemic therapy; active infection requiring systemic therapy ≤7 days prior to study drug administration, with routine antimicrobial prophylaxis permitted; positive HIV test results; patients with active hepatitis B or C (HBsAg positivity with HBV DNA titres above the upper limit of normal; HCVAb positivity with HCV RNA titres above the upper limit of normal); and persistent coronavirus (COVID-19) infection.
14. Active autoimmune disease requiring systemic treatment within the past 2 years (e.g., use of corticosteroids or immunosuppressive drugs, etc.), allowing for related replacement therapy (e.g., thyroxine, insulin, or physiological corticosteroid replacement for adrenal or pituitary insufficiency);
15. Other malignancy within 5 years prior to signing the Informed Consent Form (with the exception of non-melanoma skin cancer, cervical carcinoma in situ, limited prostate cancer, stage I endometrial cancer, or other tumours that have been effectively treated and are considered to have been cured);
16. Hypersensitivity reactions or delayed hypersensitivity reactions to certain components of vedicilizumab, patulizumab and treprostinil or similar drugs are known;
17. A concomitant disease that, in the judgement of the investigator, is a serious hazard to the safety of the subject or interferes with the subject's ability to complete the clinical study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate (ypT0/is ypN0) | 1 month after surgery
  Pathological complete response rate after neoadjuvant ( both breast and axillary lymph nodes, in which the breast may have residual carcinoma in situ);

SECONDARY OUTCOMES:
Objective remission rate (ORR) | Up to approximately 2 years
  Objective response rate.ORR assessed according to the evaluation criteria for the efficacy of solid tumors (RECIST 1.1)
Disease free survival（DFS） | Up to approximately 5 years
  From the date of surgery to the first local, regional, contralateral or distant recurrence, and death from any cause including 3- and 5-year event-free survival
Event free survival (EFS) | Up to approximately 5 years
  The time from random assignment to disease progression, including local progression before surgery; disease recurrence-local, regional, distant, ipsilateral noninvasive, or contralateral (invasive or noninvasive)-or death from any cause;
Overall survival (OS) | Date of randomization to date of death due to any cause, up to 5 years after the last subject randomized
  OS is defined as the time from the date of randomisation until the date of death due to any cause.
Adverse events | Up to approximately 2 months after surgery
  To evaluate safety including adverse event rate and adverse event grade
Change in cluster of differentiation 8 (CD8) | At baseline to surgery
  CD8 in tumor samples by biopsy at baseline and by surgery immediately after surgery would be evaluated by HE or immune staining.
Health-related quality of life - EORTC-QLQ-C30 | Up to approximately 2 years
  Change from baseline in the physical functioning subscale of the European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) scores. Scale scores range from 0-100. For functioning and global health status/ QoL scales, higher scores indicate better functioning or global health status/QoL. For symptom scales, higher scores indicate greater symptom burden
Residual cancer burden score | 1 month after surgery
  According to the extent of the residual cancer in the primary breast cancer site (mm*mm), the residual cancer (mm*mm), cell density of residual cancer (%), proportion of carcinoma in situ (%), number of positive lymph nodes and maximum diameter of lymph node metastasis (mm), the RCB index and corresponding RCB classification can be obtained. The RCB index and the corresponding RCB grade can be obtained based on the maximum diameter of the cancer (mm).
Change in tumor-infiltrating lymphocytes (TILs) | At baseline to surgery
  Defined as infiltrating lymphocytes isolated from tumor tissue.TILs in tumor samples by biopsy right before the first neoadjuvant therapy (baseline) and by surgery immediately after surgery would be evaluated by HE or immune staining。
Change in programmed cell death protein L1 (PD-L1) | At baseline to surgery
  PD1 in tumor samples by biopsy at baseline and by surgery immediately after surgery would be evaluated by HE or immune staining.

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Fang, Ph.D, Study Director — RemeGen Co., Ltd.
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No